CLINICAL TRIAL: NCT02900287
Title: Survie Des Personnes Atteintes de Cancer à la Réunion, 1998-2008 (SUCRE)
Brief Title: Cancer Survival in Reunion Island , 1998-2008 (SUCRE)
Acronym: SUCRE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/CHU/05
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Neoplasms
Keywords: Survival; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cancer survival is important to determine prognostic of patients and evaluate care and prevention health strategies. Sucre is the first study to describe cancer survival in Reunion Island. Sucre aims at evaluating five year cancer prognostic in Reunion Island by cancer site and gender. Sucre is a retrospective cohort study of cancer diagnosed between 01/01/1998 and 31/12/2008.

DETAILED DESCRIPTION:
Data are extracted from Reunion Island Cancer Registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients domiciled in Reunion Island at diagnosis
* Patients with at least 15 years of age at diagnosis
* Patients with cancer diagnosis between 01/01/1998 and 31/12/2008

Exclusion Criteria:

* Cutaneous malignant cancer expected melanoma

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population extracted from Reunion Island Cancer Registry
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
5 years related survival rate by cancer site and gender | 5 years

SECONDARY OUTCOMES:
1, 3, 5 and 10 years related survival rate by cancer site and gender | 1, 3, 5 and 10 years
1, 3, 5 and 10 years standardised survival rate by cancer site and gender | 1, 3, 5 and 10 years
1, 3, 5 and 10 years related survival rate by age at diagnosis | 1, 3, 5 and 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de La Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No